CLINICAL TRIAL: NCT02131922
Title: Study of the Effects of Intensive Treatment of Periodontitis on Blood Pressure Control and Vascular Function
Brief Title: Study of the Effects of Intensive Treatment of Periodontitis on Blood Pressure Control
Acronym: PerioBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Guzik, Prof. dr hab. med., Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOMT-01A
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Periodontitis; Hypertension
MeSH Terms: conditions — Periodontitis; Hypertension | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hygenization Treatment (Placebo Comparator): Basic oral hygiene instructions Supragingival plaque removal
  Interventions: Procedure: Dental Hygienization Treatment
- Intensive Treatment (Experimental): One-Stage Full-Mouth Disinfection. Scaling and root planing, four quadrants in one session. Extraction of radix relicta. Subgingival chlorhexidine (PerioKIN) (0.2%) in all pockets. Oral hygiene instructions.
  Interventions: Procedure: Intensive Treatment; Drug: Chlorhexidine (Intensive Treatment)

INTERVENTIONS:
Procedure: Intensive Treatment — Intensive Surgical Treatment of Periodontitis
  Other Names: Intensive Surgical Treatment of Periodontitis
  Arms: Intensive Treatment
Procedure: Dental Hygienization Treatment
  Arms: Hygenization Treatment
Drug: Chlorhexidine (Intensive Treatment) — Chlorhexidine (PerioKIN) (0.2%) implantation in dental pockets
  Arms: Intensive Treatment

SUMMARY:
Hypertensive patients with chronic periodontitis will be randomized to either intensive treatment or supragingival hygienic treatment and the effects on blood pressure will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis with three or more periodontal pockets with a probing depth (PD) > 5mm
* Bleeding of these periodontal pockets on probing
* Have at least 20 natural teeth
* Provide informed consent and willingness to cooperate with the study protocol
* Age >25 years old
* Absence of other significant oral infections.
* Primary Hypertension on stable treatment

Exclusion Criteria:

* Clinical symptoms of acute inflammatory disorders incl flu, rhinitis, sinusitis etc. within past 3 weeks
* Hospitalization for any reason within the past 3 months; Life expectancy of < 3 years;
* Allergic disorders; History of chronic infectious disease, Chronic Obstructive Pulmonary Disease (COPD), tuberculosis; chronic hepatitis B or C infection; interstitial pneumonitis, bronchiectasis; known chronic pericardial effusion, pleural effusion, or ascites; liver disease;
* Other known chronic inflammatory or autoimmune condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease
* Secondary hypertension (known plasma renin screening, abdominal ultrasound with doppler and other investigations)
* Non-basal cell malignancy or treated myelo or lymphoproliferative disease within the past 5 years;
* Known HIV positive; Immunizations within past 3 months
* Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Primary pulmonary hypertension.
* Use of systemic or local steroids or immunosuppressive agents within 6 months of the inclusion.
* Individual is pregnant or nursing
* History of alcohol abuse or unwillingness to limit alcohol consumption to less than 4 drinks per week

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Change | 3 months
  Ambulatory Blood Pressure Monitoring

SECONDARY OUTCOMES:
Flow Mediated Dilatation | 3 months
  Vascular Function Measurement

OTHER OUTCOMES:
Leukocyte Immunophenotype and Cytokine measurement | 3 months
Periodontal Health Score - Probing Depth | 3 months
Periodontal Health Score - CAL - Clinical Attachment Loss | 3 months
The Community Periodontal Index of Treatment Needs Index | 3 months
Gingival Index | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - J. Dietl Hospital, Department of Internal and Agricultural Medicine, Jagiellonian University, Krakow
  - Jagiellonian University Dental Clinic, Krakow

REFERENCES:
- [Derived] Czesnikiewicz-Guzik M, Osmenda G, Siedlinski M, Nosalski R, Pelka P, Nowakowski D, Wilk G, Mikolajczyk TP, Schramm-Luc A, Furtak A, Matusik P, Koziol J, Drozdz M, Munoz-Aguilera E, Tomaszewski M, Evangelou E, Caulfield M, Grodzicki T, D'Aiuto F, Guzik TJ. Causal association between periodontitis and hypertension: evidence from Mendelian randomization and a randomized controlled trial of non-surgical periodontal therapy. Eur Heart J. 2019 Nov 1;40(42):3459-3470. doi: 10.1093/eurheartj/ehz646. PMID 31504461